CLINICAL TRIAL: NCT02801669
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study of DU-176b in Patients With NVAF Aged 80 Years or Older Who Are Ineligible for Available Oral Anticoagulation Therapy
Brief Title: Study of DU-176b Aged 80 Years or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DU176b-C-J316; 163266 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulants; DU-176b; edoxaban; factor Xa; oral; prevention; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DU-176b 15 mg group (Experimental): DU-176b orally administered at a dose of 15 mg once daily.
  Interventions: Drug: Du-176b
- Placebo group (Placebo Comparator): Placebo orally administered once daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Du-176b — DU-176b orally administered at a dose of 15 mg once daily.
  Other Names: edoxaban
  Arms: DU-176b 15 mg group
Drug: placebo — Placebo orally administered once daily.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of edoxaban in patients with non-valvular NVAF aged 80 years or older who are ineligible for available oral anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Nonvalvular Atrial Fibrillation (NVAF) aged 80 years or older who are ineligible for available oral anticoagulation therapy

Exclusion Criteria:

* Patients with active bleeding
* Patients who have poorly controlled hypertension
* Patients who have liver dysfunction accompanied with disorder of blood coagulation

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 984 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (164):
- Japan (164):
  - Social Corporation Keigakukai Minamiosaka Hospital, Osaka, Osaka
  - Hakujikai Memorial Hospital, Adachi-ku
  - Ageo Central General Hospital, Ageo
  - Medical Corporation Aijinkai Akashi Medical Center, Akashi
  - Ako City Hospital, Akō
  - Amagasaki New Town Hospital, Amagasaki
  - Anjo Kosei Hospital, Anjo
  - Shin-Ai Kai Honda Hospital, Annaka
  - Toyooka Chuo Hospital, Asahikawa
  - Tokyo Medical and Dental University Medical Hospital, Bunkyō City
  - Nippon Medical School Hospital, Bunkyō City
  - Fukuokaken Saiseikai Futsukaichi Hospital, Chikushino-shi
  - Aichi Koseiren Chita Kosei Hospital, Chita
  - Kashinoki Internal Medicine Clinic, Date
  - Medical Plaza Edogawa, Edagawa
  - Fukui General Clinic, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Onga Nakama Medical Association Onga Hospital, Fukuoka
  - Fukushima Daiichi Hospital, Fukushima
  - Funabashi Municipal Medical Center, Funabashi
  - Gifu Heart Center, Gifu
  - Minamino Cardiovascular Hospital, Hachiōji
  - Tokyo Tenshi Hospital, Hachiōji
  - Social welfare corporation Hakodate koseiin Hakodate Goryoukaku Hospital, Hakodate
  - National Hospital Organization Hakodate Hospital, Hakodate
  - National Hospital Organization Hamada Medical Center, Hamada
  - Hamamatsu Medical Center, Hamamatsu
  - Okitama Public General Hospital, Higashinakama
  - Social Medical Corporation, the Yamatokai Foundation Central Clinic affiliated clinic of Higashiyamato Hospital, Higashiyamato
  - Hikone Municipal Hospital, Hikone
  - Kanazawa Medical University Himi Municipal Hospital, Himi
  - Hiratsuka kyosai Hospital, Hiratsuka
  - Hirosaki Stroke and Rehabilitation Center, Hirosaki
  - Local Independent Administrative Corporation Hiroshima City Hospital Organization Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Hospital Organization Mito Medical Center, Ibaraki
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Tokai University Hospital, Isehara
  - Kubo Clinic, Isesaki
  - Shimane University Hospital, Izumo
  - National Hospital Organization Kagoshima Medical Center, Kagoshima
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Kasugai Municipal Hospital, Kasugai
  - Asano Kanamachi Clinic, Katsushikachō
  - Saiseikai Kawaguchi General Hospital, Kawaguchi
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Kitasato University Medical Center, Kitamoto
  - Kobe Rosai Hospital, Kobe
  - Nose Hospital, Kobe
  - Medical Corporation Sakurakai Takahashi Hospital, Kobe
  - Nakayama Clinic of Internal Medicine and Cardiology, Kochi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kanno Reism Heart Clinic, Kosugi-shiraishi
  - Southern Tohoku Research Institute for Neuroscience, Southern Tohoku Medical Clinic, Kōriyama
  - Hoshi General Hospital, Kōriyama
  - Showa University Koto Toyosu Hospital, Kōtoku
  - Koto Hospital, Kōtoku
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kure Kyosai Hospital, Kure
  - Tanushimaru Central Hospital, Kurume
  - Kusatsu General Hospital, Kusatsu
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Machida Municipal Hospital, Machida
  - National Hospital Organization Maizuru Medical Center, Maizuru
  - New Tokyo Heart Clinic, Matsudo
  - Matsue City Hospital, Matsue
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Miyazaki Medical Association Hospital, Miyazaki
  - University of Miyazaki Hospital, Miyazaki
  - Iwate Prefectural Central Hospital, Morioka
  - Nagasaki Harbor Medical Center, Nagasaki
  - Nagoya Ekisaikai Hospital, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Ohama Daiichi Hospital, Naha
  - Naha City Hospital, Naha
  - Takanohara Central Hospital, Nara
  - JCHO Nihonmatsu Hospital, Nihonmatsu
  - Meiwa Hospital, Nishinomiya
  - Ohyama Memorial Hospital, Nishiwaki
  - Ogawa Cardiovascular Internal Medicine Clinic, Obihiro
  - Shimada Hospital, Ogōri-shimogō
  - Sakurabashi Watanabe Hospital, Osaka
  - Osaka City Juso Hospital, Osaka
  - Kitada Clinic, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - National Hospital Organization Osaka Minami Medical Center, Osaka
  - Sato Hospital, Osaka
  - Otaru Kyokai Hospital, Otaru
  - Ogaki Municipal Hospital, Ōgaki
  - Oita Prefectural Hospital, Ōita
  - Kouhoukai Takagi Hospital, Ōkawa
  - Ome Municipal General Hospital, Ōme
  - Omihachiman Community Medical Center, Ōmihachiman
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Omori Sanno Hospital, Ōta-ku
  - JCHO Shiga Hospital, Ōtsu
  - Saga-Ken Medical Centre Koseikan, Saga
  - Saitama City Hospital, Saitama
  - Saitama Memorial Hospital, Saitama
  - Saku Central Hospital Advanced Care Center, Saku
  - Kin-ikyo Chuo Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - National Hospital Organization Hokkaido Medical Center, Sapporo
  - Sapporo Nishimaruyama Hospital, Sapporo
  - Miyanomori Memorial Hospital, Sapporo
  - Hokkaido Cardiovascular Hospital, Sapporo
  - Shukokai Internal Medicine Sato Hospital, Sendai
  - KKR Tohoku Kosai Hospital, Sendai
  - National Hospital Organization Sendai Medical Center, Sendai
  - Tosei General Hospital, Seto
  - National Hospital Organization Kanmon Medical Center, Shimonoseki
  - Dokkyo Medical University Hospital, Shimosuga
  - Tokyo Heart Center, Shinagawa-Ku
  - Showa University Hospital, Shinagawa-Ku
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku
  - Shirakawa Hospital, Shirakawa
  - Iwate Medical University Hospital, Shiwa-gun
  - National Hospital Organization Shizuoka Medical Center, Shizuoka
  - Ikeda Kinen Hospital, Sukagawa
  - Iwase General Hospital, Sukagawa
  - Hyogo Prefectural Awaji Medical Center, Sumoto
  - Nagano Prefectural Shinshu Medical Hospital, Suzaka
  - National Hospital Organization Disaster Medical Center, Tachikawa
  - Social Insurance Tagawa Hospital, Tagawa
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Kouseiren Takaoka Hospital, Takaoka
  - Medical Corporation Aishinkai Higashi Takarazuka Satoh Hospital, Takarazuka
  - Kan-etsu Chu-oh Hospital, Takasaki
  - Takatsuki General Hospital, Takatsuki
  - National Hospital Organization Minami Wakayama Medical Center, Tanabe
  - Tenri Hospital, Tenri
  - Kuwanomi Hongou Clinic, Tokorozawa
  - Saino Clinic, Tokorozawa
  - Tokorozawa Heart Center, Tokorozawa
  - Tokushima University Hospital, Tokushima
  - Tokushima Prefectural Central Hospital, Tokushima
  - Nerima General Hospital, Tokyo
  - Tomakomai City Hospital, Tomakomai
  - Public Tomioka General Hospital, Tomioka
  - Yamaguchi Clinic, Toshima-ku
  - Yayoigaoka Kage Hospital, Tosu
  - National Hospital Organization Toyohashi Medical Center, Toyohashi
  - TOYOTA Memorial Hospital, Toyota
  - National Hospital Organization Ehime Medical Center, Tōon
  - Tsukuba Memorial Hospital, Tsukuba
  - Okinawa Prefectural Chubu Hospital, Uruma
  - National Hospital Organization Tochigi Medical Center, Utsunomiya
  - Uwajima City Hospital, Uwajima
  - Wakayama Rosai Hospital, Wakayama
  - Nagata Hospital, Yanagawa
  - Kumamoto General Hospital, Yatsushiro
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Yokohama Rosai Hospital, Yokohama
  - Showa University Fujigaoka Hospital, Yokohama
  - JCHO Yokohama Chuo Hospital, Yokohama
  - Yokohama City Minato Red Cross Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama
  - Yokohama Minami Kyousai Hospital, Yokohama
  - National Hospital Organization Yokohama Medical Center, Yokohama
  - Yokohama Sakae Kyosai Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Akao M, Yamashita T, Fukuzawa M, Hayashi T, Okumura K. Efficacy and Safety of Low-Dose Edoxaban by Body Weight in Very Elderly Patients With Atrial Fibrillation: A Subanalysis of the Randomized ELDERCARE-AF Trial. J Am Heart Assoc. 2024 Feb 6;13(3):e031506. doi: 10.1161/JAHA.123.031506. Epub 2024 Jan 19. PMID 38240204
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Mikami T, Hirabayashi K, Okawa K, Betsuyaku T, Watanabe S, Imamura Y, Tanizawa K, Hayashi T, Akao M, Yamashita T, Okumura K. Laboratory Test Predictors for Major Bleeding in Elderly (>/=80 Years) Patients With Nonvalvular Atrial Fibrillation Treated With Edoxaban 15 mg: Sub-Analysis of the ELDERCARE-AF Trial. J Am Heart Assoc. 2022 Sep 6;11(17):e024970. doi: 10.1161/JAHA.122.024970. Epub 2022 Sep 3. PMID 36056729
- [Derived] Kuroda M, Tamiya E, Nose T, Ogimoto A, Taura J, Imamura Y, Fukuzawa M, Hayashi T, Akao M, Yamashita T, Lip GYH, Okumura K. Effect of 15-mg Edoxaban on Clinical Outcomes in 3 Age Strata in Older Patients With Atrial Fibrillation: A Prespecified Subanalysis of the ELDERCARE-AF Randomized Clinical Trial. JAMA Cardiol. 2022 Jun 1;7(6):583-590. doi: 10.1001/jamacardio.2022.0480. PMID 35416910
- [Derived] Yoshida T, Nakamura A, Funada J, Amino M, Shimizu W, Fukuzawa M, Watanabe S, Hayashi T, Yamashita T, Okumura K, Akao M. Efficacy and Safety of Edoxaban 15 mg According to Renal Function in Very Elderly Patients With Atrial Fibrillation: A Subanalysis of the ELDERCARE-AF Trial. Circulation. 2022 Mar;145(9):718-720. doi: 10.1161/CIRCULATIONAHA.121.057190. Epub 2022 Feb 28. No abstract available. PMID 35226559
- [Derived] Okumura K, Akao M, Yoshida T, Kawata M, Okazaki O, Akashi S, Eshima K, Tanizawa K, Fukuzawa M, Hayashi T, Akishita M, Lip GYH, Yamashita T; ELDERCARE-AF Committees and Investigators. Low-Dose Edoxaban in Very Elderly Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 29;383(18):1735-1745. doi: 10.1056/NEJMoa2012883. Epub 2020 Aug 30. PMID 32865374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 984 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment at 164 clinic centers in Japan. Of the 984 participants, 982 received treatment.
Pre-assignment Details: Participants were assigned to the DU-176b or placebo group in a 1:1 ratio using a stratified randomization method with the CHADS2 index score (≤2, ≥3) as a stratification factor.
Groups:
- DU-176b 15 mg: Participants who were randomized to oral DU-176b administered at a dose of 15 mg once daily.
- Placebo: Participants who were randomized to oral placebo administered once daily.
Period: Overall Study
Arm/Group | DU-176b 15 mg | Placebo
Started | 492 | 492
Received at Least 1 Dose of Study Drug | 492 | 490
Completed | 341 | 340
Not Completed | 151 | 152
Not completed — Death | 66 | 69
Not completed — Withdrawal by Subject | 81 | 77
Not completed — Other | 4 | 6

BASELINE CHARACTERISTICS:
Population: Baseline demographics were assessed in the intent-to-treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b 15 mg | Placebo | Total
Number analyzed (Participants) | 492 | 492 | 984
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.7 (4.22) | 86.4 (4.27) | 86.6 (4.24)
Age, Customized [Count of Participants; unit: Participants]
  <85 years | 173 | 181 | 354
  85 to <90 years | 190 | 184 | 374
  90 to <95 years | 110 | 106 | 216
  95 years or older | 19 | 21 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 285 | 565
  Male | 212 | 207 | 419
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 492 | 492 | 984
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 492 | 492 | 984

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Endpoint of Stroke and Systemic Embolic Events (SEE) in Participants Who Were Administered DU-176b Compared With Placebo
Description: Stroke was defined as an abrupt onset, over minutes to hours, of symptoms representing focal neurological deficit in the domain supplied by a single brain artery (including the retinal artery) and that was not due to an identifiable non-vascular cause (such as brain tumor or trauma). The deficit symptoms had to either last for more than 24 hours or result in death within 24 hours of symptom onset.
  A systemic embolic event (SEE) was defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms (eg, atherosclerosis and instrumentation).
Time Frame: Randomization up to the time of onset of the initial composite event of stroke or systemic embolic event, or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: The primary outcome was assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 15 | 44
Statistical Analysis 1: Comparison: DU-176b 15 mg vs Placebo; This statistical analysis assesses the annual incidence of composite event of stroke and SEE between treatment groups; Test type: Other; p = 0.0003, Regression, Cox; The treatment groups were compared using a Cox proportional hazard model with the CHADS2 score (<= 2 or >= 3) as covariate; Cox Proportional Hazard = 0.339, 95% CI 2-sided [0.188 to 0.608]

2. Primary Outcome: Number of Participants With Stroke and Systemic Embolic Events (SEE), Including Subcomponents of Stroke and Composite Event of Ischemic Stroke and SEE in Participants Who Were Administered DU-176b Compared With Placebo
Description: Stroke was defined as an abrupt onset, over minutes to hours, of symptoms representing focal neurological deficit in the domain supplied by a single brain artery (including the retinal artery) and that was not due to an identifiable non-vascular cause (such as brain tumor or trauma). The deficit symptoms had to either last for more than 24 hours or result in death within 24 hours of symptom onset. Subcomponents of stroke (ischemic and hemorrhagic) were also reported.
  A systemic embolic event (SEE) was defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms (eg, atherosclerosis and instrumentation).
Time Frame: as for outcome 1
Population: The primary outcome was assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants
  Stroke | 12 | 40
  Systemic Embolic Events (SEE) | 3 | 6
  Ischaemic Stroke | 12 | 39
  Hemorrhagic Stroke | 0 | 2
  Ischemic Stroke/SEE | 15 | 43
Statistical Analysis 1: Comparison: DU-176b 15 mg vs Placebo; This statistical analysis assesses the annual incidence of stroke between treatment groups; Test type: Other; Cox Proportional Hazard = 0.299, 95% CI 2-sided [0.157 to 0.570] — The treatment groups were compared using a Cox proportional hazard model with the CHADS2 score (<= 2 or >= 3) as covariate
Statistical Analysis 2: Comparison: DU-176b 15 mg vs Placebo; This statistical analysis assesses the annual incidence of SEE between treatment groups; Test type: Other; Cox Proportional Hazard = 0.503, 95% CI 2-sided [0.126 to 2.011] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: DU-176b 15 mg vs Placebo; This statistical analysis assesses the annual incidence of ischemic stroke between treatment groups; Test type: Other; Cox Proportional Hazard = 0.306, 95% CI 2-sided [0.160 to 0.585] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: DU-176b 15 mg vs Placebo; This statistical analysis assesses the annual incidence of ischemic stroke/SEE between treatment groups; Test type: Other; Cox Proportional Hazard = 0.347, 95% CI 2-sided [0.193 to 0.624] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants With a Composite Endpoint of Stroke, Systemic Embolic Events (SEE), and Death Due to Cardiovascular in Participants Who Were Administered DU-176b Compared With Placebo
Description: as for outcome 1
Time Frame: Randomization up to the time of onset of the initial composite event of stroke, systemic embolic event, or death due to CV, or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Secondary outcomes were assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 52 | 72

4. Secondary Outcome: Number of Participants With a Composite Endpoint of a Major Adverse Cardiovascular Event (MACE) in Participants Who Were Administered DU-176b Compared With Placebo
Description: Major adverse cardiovascular events (MACE) included a composite of non-fatal myocardial infarction (MI), non-fatal stroke, non-fatal systemic embolic events (SEE), and deaths due to cardiovascular (CV) or bleeding.
  Stroke was defined as an abrupt onset, over minutes to hours, of symptoms representing focal neurological deficit in the domain supplied by a single brain artery (including the retinal artery) and that was not due to an identifiable non-vascular cause (such as brain tumor or trauma). The deficit symptoms had to either last for more than 24 hours or result in death within 24 hours of symptom onset.
  A SEE was defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms (eg, atherosclerosis and instrumentation).
Time Frame: Randomization up to the time of onset of the initial MACE event, or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Secondary outcomes were assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 51 | 72

5. Secondary Outcome: Number of Participants With a Composite Endpoint of Stroke, Systemic Embolic Events (SEE), and All-Cause Mortality in Participants Who Were Administered DU-176b Compared With Placebo
Description: Stroke was defined as an abrupt onset, over minutes to hours, of symptoms representing focal neurological deficit in the domain supplied by a single brain artery (including the retinal artery) and that was not due to an identifiable non-vascular cause (such as brain tumor or trauma). The deficit symptoms had to either last for more than 24 hours or result in death within 24 hours of symptom onset.
  A systemic embolic event (SEE) was defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms (eg, atherosclerosis and instrumentation).
  All-cause mortality was defined as death due to cardiovascular and mortality due to all other causes.
Time Frame: Randomization up to the time of onset of the initial composite event of stroke, SEE, all-cause mortality, or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Secondary outcomes were assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 74 | 98

6. Secondary Outcome: Number of Participants With Net Clinical Benefit in Participants Who Were Administered DU-176b Compared With Placebo
Description: Net clinical benefit included a composite of stroke, systemic embolic events (SEE), major bleeding, and all-cause mortality. Stroke was defined as an abrupt onset of symptoms representing focal neurological deficit in the domain supplied by a single brain artery that was not due to an identifiable non-vascular cause. The deficit symptoms had to either last >24 hours or result in death within 24 hours of symptom onset. A SEE was defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms. Major bleeding was defined as overt bleeding that met at least 1 of the following criteria: fatal bleeding; retroperitoneal, intracranial, intraocular, intrathecal, intraarticular, or pericardial bleeding, or symptomatic intramuscular bleeding accompanied by compartment syndrome; or clinically overt bleeding that decreased hemoglobin by at least 2.0 g/dL and required blood transfusion.
Time Frame: Randomization up to the time of onset of the initial composite event of stroke, SEE, major bleeding, all-cause mortality, or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Secondary outcomes were assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 87 | 103

7. Secondary Outcome: Number of Participants With All-Cause Mortality in Participants Who Were Administered DU-176b Compared With Placebo
Description: All-cause mortality was defined as death due to cardiovascular and mortality due to all other causes.
Time Frame: Randomization up to death (due to any cause), or study discontinuation, or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Secondary outcomes were assessed in the Intent-to-Treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 492
Participants | 66 | 69

8. Secondary Outcome: Number of Participants With Major Bleeding During On-Treatment Period in Participants Who Were Administered DU-176b Compared With Placebo
Description: Major bleeding was defined as overt bleeding that met at least 1 of the following criteria: fatal bleeding; retroperitoneal, intracranial, intraocular, intrathecal, intraarticular, or pericardial bleeding, or symptomatic intramuscular bleeding accompanied by compartment syndrome; or clinically overt bleeding that decreased hemoglobin by at least 2.0 g/dL and required blood transfusion.
Time Frame: Baseline up to study discontinuation or end of study (whichever comes first), up to 3 years 2 months postdose (maximum follow-up time)
Population: Safety outcomes were assessed in the Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 490
Participants
  Major bleeding | 20 | 11
  Major bleeding, Intracranial haemorrhage | 2 | 4
  Fatal bleeding | 0 | 2
  Fatal bleeding, Intracranial haemorrhage | 0 | 1
  Fatal bleeding, Non-Intracranial haemorrhage | 0 | 1
  Life-threatening bleeding | 8 | 4

9. Secondary Outcome: Number of Participants With Major Bleeding or Clinically Relevant Non-major Bleedings During On-Treatment Period in Participants Who Were Administered DU-176b Compared With Placebo
Description: Major bleeding was defined as overt bleeding that met at least 1 of the following criteria: fatal bleeding; retroperitoneal, intracranial, intraocular, intrathecal, intraarticular, or pericardial bleeding, or symptomatic intramuscular bleeding accompanied by compartment syndrome; or clinically overt bleeding that decreased hemoglobin by at least 2.0 g/dL and required blood transfusion. Clinically overt bleeding that required treatment was taken to be clinically relevant non-major bleeding, including for example (but was not limited to) the bleeding that led to the diagnostic tests and treatments as specified in the protocol. The clinically overt bleeding requiring treatment did not include outpatient examinations that did not involve any of the medical procedures (diagnostic tests or treatments) as specified in the protocol.
Time Frame: as for outcome 8
Population: Safety outcomes were assessed in the Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 490
Participants
  Major or clinically relevant non-major bleeding | 97 | 62
  Clinically relevant non-major bleeding | 81 | 52

10. Secondary Outcome: Number of Participants With All Bleeding Events and Minor Bleeding Events During On-Treatment Period in Participants Who Were Administered DU-176b Compared With Placebo
Description: All bleeding events include major and clinically relevant non-major bleeding events.
  Other overt bleeding events that did not meet the criteria for major bleeding or clinically relevant non-major bleeding were taken to be minor bleeding (for example, epistaxis that did not require treatment). All events other than the above (such as a decrease in hemoglobin without overt bleeding) were classified as "non-bleeding event."
Time Frame: as for outcome 8
Population: Safety outcomes were assessed in the Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | DU-176b 15 mg | Placebo
Number analyzed (Participants) | 492 | 490
Participants
  All bleeding | 241 | 202
  Minor bleeding | 190 | 177

11. Secondary Outcome: Plasma Concentration of DU-176 in Participants Who Were Administered DU-176b
Time Frame: Week 8: Predose,1-3 hours (h) and 4-8 h postdose
Population: Plasma concentration was assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DU-176b 15 mg
Number analyzed (Participants) | 451
ng/mL
  Week 8: Predose (trough): number analyzed (Participants) | 427
  Week 8: Predose (trough) | 17.3 (13.9)
  Week 8: 1-3 h: number analyzed (Participants) | 447
  Week 8: 1-3 h | 93.3 (57.8)
  Week 8: 4-8 h: number analyzed (Participants) | 125
  Week 8: 4-8 h | 93.4 (37.5)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 3 years 2 months postdose.
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event that first appears during treatment, which is absent before treatment or which worsens relative to pre-treatment state. TEAEs are reported in the Safety Analysis Set.
Arm/Group | DU-176b 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 66/492 | 69/490
Serious Adverse Events (participants affected / at risk) | 220/492 | 238/490
Other Adverse Events (participants affected / at risk) | 461/492 | 454/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DU-176b 15 mg (N=492) | Placebo (N=490)
Pyelonephritis acute (Infections and infestations) | 1 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Infections and infestations) | 26 | 34
Urinary tract infection (Infections and infestations) | 5 | 7
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Dehydration (Metabolism and nutrition disorders) | 14 | 10
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Cerebral infarction (Nervous system disorders) | 3 | 18
Embolic stroke (Nervous system disorders) | 3 | 10
Cataract (Eye disorders) | 5 | 6
Cardiac failure congestive (Cardiac disorders) | 31 | 28
Cardiac failure (Cardiac disorders) | 25 | 30
Cardiac failure chronic (Cardiac disorders) | 14 | 6
Cardiac failure acute (Cardiac disorders) | 7 | 4
Sinus node dysfunction (Cardiac disorders) | 2 | 5
Acute myocardial infarction (Cardiac disorders) | 0 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Femur fracture (Injury, poisoning and procedural complications) | 9 | 15
Spinal compression fracture (Injury, poisoning and procedural complications) | 7 | 13
Bronchitis (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 2
Periodontitis (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 1 | 3
Bacteraemia (Infections and infestations) | 3 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Marasmus (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 3
Loss of consciousness (Nervous system disorders) | 4 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 2
Cerebellar infarction (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 1
Lacunar infarction (Nervous system disorders) | 1 | 2
Dementia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 2 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4
Ventricular fibrillation (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 3 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Large intestine polyp (Gastrointestinal disorders) | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dumping syndrome (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 4
Bile duct stone (Hepatobiliary disorders) | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Crowned dens syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Renal impairment (Renal and urinary disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Disuse syndrome (General disorders) | 3 | 3
Pyrexia (General disorders) | 4 | 1
Chest pain (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 4
Rib fracture (Injury, poisoning and procedural complications) | 3 | 1
Heat illness (Injury, poisoning and procedural complications) | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Removal of foreign body from joint (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DU-176b 15 mg (N=492) | Placebo (N=490)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 42 | 16
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 73 | 88
Haematuria (Renal and urinary disorders) | 44 | 14
Nasopharyngitis (Infections and infestations) | 111 | 121
Pneumonia (Infections and infestations) | 47 | 53
Urinary tract infection (Infections and infestations) | 27 | 27
Bronchitis (Infections and infestations) | 35 | 18
Anaemia (Blood and lymphatic system disorders) | 39 | 21
Dehydration (Metabolism and nutrition disorders) | 37 | 32
Cardiac failure congestive (Cardiac disorders) | 42 | 51
Hypertension (Vascular disorders) | 26 | 20
Constipation (Gastrointestinal disorders) | 52 | 45
Diarrhoea (Gastrointestinal disorders) | 34 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 31
Contusion (Injury, poisoning and procedural complications) | 43 | 49
Cardiac failure (Cardiac disorders) | 45 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT02801669/Prot_SAP_000.pdf